CLINICAL TRIAL: NCT03365349
Title: Comparison Between Two Narrative Medicine Approaches in Type 1 Diabetes (T1D): a Prospective Randomized Study
Brief Title: Two Narrative Medicine Interventions in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Agnes Hartemann, head of the diabetes department at the university hospital Pitié Salpetrière Paris, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDV
Record Dates: First submitted 2017-11-17; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Type1diabetes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- living theatre (Experimental): One session consisting for the patient of telling a story about his/her own life with diabetes , which is first written and then transformed to a script to be played by professional actors co-directed by the patient with the support of the Director to create a little play.
  Interventions: Other: participating in a session of "living theatre"
- writing workshop (Active Comparator): one session consisting for the patient of writing a "Letter to his/her own diabetes" and then to read it to the group of patients and the healthcare providers.
  Interventions: Other: writing workshop

INTERVENTIONS:
Other: participating in a session of "living theatre" — participating to a session of "living theatre" which consists in writing a story about life with diabetes, which is then transformed to a script to be played by professional actors co-directed by the patient with the support of the Director to create a short play
  Arms: living theatre
Other: writing workshop — one session consisting for the patient of writing a "Letter to his/her own diabetes" and then to read it to the group of patients and the healthcare providers.
  Arms: writing workshop

SUMMARY:
a randomized prospective study aims at comparing the impact of a "living theater" session with a simple "writing workshop " on emotional distress (Problem Areas in Diabetes Questionnaire PAID) and illness perception ( Illness Perception Questionnaire IPQR) during a 5 day education course

DETAILED DESCRIPTION:
This randomized prospective pilot study aims at comparing the impact of a "living theater" session with a simple "writing workshop " on emotional distress (Problem Areas in Diabetes Questionnaire PAID) and illness perception ( Illness Perception Questionnaire IPQR) during a 5 day education course on Functional Insulin Therapy (FIT). Questionaries at T0 (course day 1 ) and T1 (3 months later). qualitative interviews in a sub group of patients random G1 and G2 subgroup at T1, with a general inductive approach to capture all representations

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes

Exclusion Criteria:

* no french language

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-02-01; Primary Completion 2013-02-28 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline IPQR (Illness Perception Questionnaire) score at 3 months | 3 months after intervention
  Illness Perception Questionnaire (IPQR) There is no total score for IPQR Nine subscales are reported for IPQR. High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition. High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition. Minimal and maximal score are respectively 0 and 14 for identity, 0 and 30 for timeline, consequences, personal control, and emotional representations, 0 and 25 for treatment control and illness coherence illness, 0-20 for timeline cyclical

SECONDARY OUTCOMES:
comparison of the two groups concerning answers to qualitative interviews at T 3 months after the intervention | 3 months after intervention
  A psychologist conducted qualitative interviews according to a blinded process in a subgroup of 6 patients at T3 months, with a general inductive approach to capture all representations on diabetes and the session. Transcribed Interviews were analyzed regarding inductive coding and 2 independent investigators built and tested a coding schedule.

IPD SHARING:
Plan to Share IPD: No